CLINICAL TRIAL: NCT03333551
Title: A Pilot Study to Evaluate 18F Florbetapir Binding to Cardiac Amyloid in Patients Undergoing Chemotherapy
Brief Title: Cardiac Uptake of 18F Florbetapir in Patients Undergoing Chemotherapy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow recruitment.
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Christopher Mueller, MD, Assistant Professor Department of Medicine., Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 29197
Record Dates: First submitted 2017-10-13; First posted 2017-11-07 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Cardiac Amyloidosis
Keywords: AL Cardiac Amyloidosis; 18F-Florbetapir (Amyvid)
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — florbetapir

STUDY DESIGN:
Intervention Model Description: each participant will be subject to the intervention which is PET/CT imaging (Positron emission tomography-computed tomography) with florbetapir F-18
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with AL cardiac amyloid (Experimental): Patients enrolled will be patients > 18 years of age with a clinical diagnosis of cardiac AL amyloidosis (typical echocardiographic or MRI findings, NT-ProBNP levels above 332 pg/mL, cardiac or extra cardiac histological evidence of light chain amyloidosis) with plans to undergo plasma cell directed chemotherapy.
  Interventions: Drug: F18 Florbetapir (amyvid) cardiac PET/CT imaging

INTERVENTIONS:
Drug: F18 Florbetapir (amyvid) cardiac PET/CT imaging — Patients with cardiac amyloidosis (AL) undergoing planned plasma cell directed chemotherapy will have F-18 florbetapir (amyvid) cardiac PET/CT imaging prior to starting chemotherapy and six months after onset of treatment.
  Other Names: Amyvid

SUMMARY:
This is a pilot study designed to assess for relative change in cardiac 18F Florbetapir uptake in patients with AL cardiac amyloidosis after appropriate chemotherapy.

DETAILED DESCRIPTION:
Current research involving [18F]-florbetapir in relationship to cardiac amyloid has taken advantage of the ability of the radiopharmaceutical to bind specifically to amyloid fibrils. It has previously been established that the degree of radiotracer uptake correlates with the density of Beta-amyloid plaque. The ability to quantify this uptake makes [18F]-florbetapir imaging a potential tool to evaluate cardiac response in patients undergoing therapy for AL amyloidosis. It would provide a much-needed tool to monitor cardiac response to chemotherapy to potentially adjust chemotherapy if response was not adequate. It could also provide a tool by which investigators would be able to evaluate new therapies designed to decrease the burden of formed amyloid fibrils within the heart.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged > 18 years are eligible.
2. Patient must provide informed consent to participate in the study protocol.
3. All patients must have clinical diagnosis of cardiac AL amyloidosis (typical echocardiographic or cardiac MRI findings, NT-ProBNP levels above 332 pg/mL, cardiac or extra cardiac histological evidence of light chain amyloidosis).
4. Planned plasma cell-directed chemotherapy.
5. A negative pregnancy test will be required for all women of child bearing potential, breast feeding is not permitted.
6. Patients must be able to undergo PET-CT imaging
7. Patients must be able to complete 6-minute walk test

Exclusion Criteria:

1. Severe claustrophobia
2. Pregnancy
3. Allergy to F-18 florbetapir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Relative change in cardiac uptake of 18F florbetapir prior to chemotherapy and after six months of chemotherapy. | six months
  Levels of 18F florbetapir cardiac uptake at onset of chemotherapy will be compared with levels after six months of chemotherapy on repeat imaging.

SECONDARY OUTCOMES:
six minute walk test | twelve months
  Change in Distance covered on six minute walk test at onset of chemotherapy will be compared to distance covered after six months of chemotherapy Distance at onset vs six months will be correlated with changes in 18F florbetapir cardiac uptake on cardiac PET/CT imaging between 0 and 6 months. Overall change in distance walked during 6 minute walk prior to starting chemotherapy and after 12 months of chemotherapy will be compared to any changes in 18F florbetapir cardiac uptake on cardiac PET/CT imaging between 0 and 6 months.
Hematologic response | 12 months
  correlation of hematologic response to treatment at 6 months and 18F florbetapir cardiac uptake changes between 0 and 6 months. Hematologic response after 12 months will also be compared to any changes in 18F florbetapir cardiac uptake between 0 and 6 months.
Cardiac response | 12 months
  Cardiac response as defined by changes in NT proBNP (N Terminal proBNP) levels and cardiac Troponin T levels will be correlated with changes in 18F florbetapir cardiac uptake between 0 and 6 months. Changes in Cardiac troponin T and NT pro BNP levels after 12 months will also be correlated with changes in 18F florbetapir cardiac uptake between 0 and 6 months.
Patient related outcomes | 12 months
  Correlation of hematologic response to results of patient related outcomes survey completed at 0, 6, and 12 months
Patient related outcomes | 12 months
  Correlation of cardiac response to results of patient related outcomes survey completed at 0, 6, and 12 months
Patient related outcomes | 12 months
  Correlation changes in 18F florbetapir cardiac uptake between 0 and 6 months to results of patient related outcomes survey completed at 0, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Chris Mueller, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Esplin BL, Gertz MA. Current trends in diagnosis and management of cardiac amyloidosis. Curr Probl Cardiol. 2013 Feb;38(2):53-96. doi: 10.1016/j.cpcardiol.2012.11.002. PMID 23337445
- [Background] Dorbala S, Vangala D, Semer J, Strader C, Bruyere JR Jr, Di Carli MF, Moore SC, Falk RH. Imaging cardiac amyloidosis: a pilot study using (1)(8)F-florbetapir positron emission tomography. Eur J Nucl Med Mol Imaging. 2014 Sep;41(9):1652-62. doi: 10.1007/s00259-014-2787-6. Epub 2014 May 20. PMID 24841414
- [Background] Osborne DR, Acuff SN, Stuckey A, Wall JS. A Routine PET/CT Protocol with Streamlined Calculations for Assessing Cardiac Amyloidosis Using (18)F-Florbetapir. Front Cardiovasc Med. 2015 May 8;2:23. doi: 10.3389/fcvm.2015.00023. eCollection 2015. PMID 26664895
- [Background] Lister-James J, Pontecorvo MJ, Clark C, Joshi AD, Mintun MA, Zhang W, Lim N, Zhuang Z, Golding G, Choi SR, Benedum TE, Kennedy P, Hefti F, Carpenter AP, Kung HF, Skovronsky DM. Florbetapir f-18: a histopathologically validated Beta-amyloid positron emission tomography imaging agent. Semin Nucl Med. 2011 Jul;41(4):300-4. doi: 10.1053/j.semnuclmed.2011.03.001. PMID 21624563
- [Background] Park MA, Padera RF, Belanger A, Dubey S, Hwang DH, Veeranna V, Falk RH, Di Carli MF, Dorbala S. 18F-Florbetapir Binds Specifically to Myocardial Light Chain and Transthyretin Amyloid Deposits: Autoradiography Study. Circ Cardiovasc Imaging. 2015 Aug;8(8):10.1161/CIRCIMAGING.114.002954 e002954. doi: 10.1161/CIRCIMAGING.114.002954. PMID 26259579
- [Background] Sikkink LA, Ramirez-Alvarado M. Cytotoxicity of amyloidogenic immunoglobulin light chains in cell culture. Cell Death Dis. 2010 Nov 11;1(11):e98. doi: 10.1038/cddis.2010.75. PMID 21368874
- [Background] Merlini G, Bellotti V. Molecular mechanisms of amyloidosis. N Engl J Med. 2003 Aug 7;349(6):583-96. doi: 10.1056/NEJMra023144. No abstract available. PMID 12904524